CLINICAL TRIAL: NCT02126007
Title: Fatigue Management in HIV: A Sleep and Circadian Rhythm Pilot Intervention
Brief Title: Fatigue Management in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIV-fatigue
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Fatigue
Keywords: fatigue; HIV; behavioral intervention; sleep
MeSH Terms: conditions — Fatigue | interventions — Sleep; Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep and Rhythm Intervention (Experimental): This arm receives a 4-week behavioral intervention aimed at improving sleep and circadian rhythms, and thereby reducing fatigue.
  Interventions: Behavioral: Sleep and Rhythm Intervention
- Dietary Modifications (Placebo Comparator): This arm receives a 4-week placebo intervention focused on dietary modifications for reducing fatigue.
  Interventions: Behavioral: Dietary Modifications

INTERVENTIONS:
Behavioral: Sleep and Rhythm Intervention
  Arms: Sleep and Rhythm Intervention
Behavioral: Dietary Modifications
  Arms: Dietary Modifications

SUMMARY:
This randomized clinical trial (RCT) pilot study as two main objectives:

* determine the overall feasibility of a behavioral intervention for managing fatigue among older adults with HIV infection.
* to estimate effect sizes for group differences at 1, 2, and 3 months on five dimensions of fatigue.

The investigators hypothesize that adherence, satisfaction, and attrition will be similar for the active intervention group and the attention control group. The investigators also hypothesize that all five dimensions will improve in the intervention group compared to controls over time, and that Cohen's d (Standard Deviation units) will be greater than 0.5 SD units for all five fatigue dimensions at all three post-intervention time points.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HIV infection
* Be at least 50 years of age
* Have a Fatigue Severity Score13 > 4.0
* Be retired or on disability
* Be willing to wear a FitBit One Tracker and keep a 7-day diary at 4 time points (electronic, paper, or other convenient format)
* Be able to speak, understand, and read English
* Have a telephone, cell phone, computer access, or other means of communication

Exclusion Criteria:

* Current temporary, part-time, or full-time employment
* Planning to travel or be away from home during the 3-month study time frame
* Being pre- or peri-menopausal because of fluctuations in vasomotor symptoms over time
* Taking hormones to treat symptoms of menopause
* Brief Interview for Mental Status score < 13
* AIDS dementia diagnosis
* Diagnosed sleep disorder that would not be responsive to behavioral interventions (sleep apnea, restless legs, etc.).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Morning fatigue severity | 3 months
  self-report ratings of morning fatigue severity (Lee Fatigue Scale)
Evening fatigue severity | 3 months
  self-report ratings of evening fatigue severity (Lee Fatigue Scale)
Lack of energy - frequency | 3 months
  self-report rating of the frequency of a lack of energy in past week (single item from Memorial Symptom Assessment Scale)
Lack of energy - severity | 3 months
  self-report rating of the severity of a lack of energy in past week (single item from Memorial Symptom Assessment Scale)
Lack of energy - distress | 3 months
  self-report rating of the distress due to a lack of energy in past week (single item from Memorial Symptom Assessment Scale)
Attrition | 3 months
  Proportion of participants who do not complete the study
Satisfaction with the intervention | 3 months
  Ratings of participant satisfaction with the 6 intervention components
Adherence to intervention | 3 months
  Self-reported adherence to each of the 6 behavioral intervention components

SECONDARY OUTCOMES:
Objectively measured sleep duration | 3 months
  Mean night-time sleep duration in minutes during the 7-day assessment period as estimated by FitBit monitor.
Objectively measured sleep quality | 3 months
  Mean number of night-time wakes during the 7-day assessment period as estimated by FitBit monitor.
Objectively-measured activity | 3 months
  Mean number of daily steps during 7-day assessment period
Sleep medication use | 3 months
  Self-reported use of sleep medication during the 7-day assessment period
Self-reported sleep quality | 3 months
  Pittsburgh Sleep Quality Index (PSQI) total score
Depressed mood | 3 months
  Hospital Anxiety and Depression Scale (HADS) - depression subscore
Anxious mood | 3 months
  Hospital Anxiety and Depression Scale (HADS) - anxiety subscore
Physical function | 3 months
  Short Form (SF)-36 physical function score
Cognitive function | 3 months
  SF-36 cognitive function score
Medication adherence | 3 months
  AIDS Clinical Trials Group (ACTG) Adherence score
Daytime sleepiness | 3 months
  Epworth Sleepiness Scale (ESS) - total score
Fatigue interference with daytime function | 3 months
  Fatigue Severity Scale - mean score
Sleep behavior | 3 months
  Sleep Behavior Self-Rating Scale (SBSRS) - total score

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Lee, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Lee KA, Jong S, Gay CL. Fatigue management for adults living with HIV: A randomized controlled pilot study. Res Nurs Health. 2020 Jan;43(1):56-67. doi: 10.1002/nur.21987. Epub 2019 Oct 14. PMID 31612533